CLINICAL TRIAL: NCT06721858
Title: Effects of Emotion-Focused Therapy (EFT) on Mood Awareness and Emotional Reactivity in Bipolar Patients
Brief Title: Effects of Emotion-Focused Therapy (EFT) on Mood Awareness and Emotional Reactivity in Bipolar PatientsAwareness and Emotional Reactivity
Acronym: EFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Gullu Yazkan, PhD, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-KAEK-23/ 49
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Therapy, Directly Observed
Keywords: emotion focused therapy; emotional reactivity; mood awareness; bipolar disorder
MeSH Terms: conditions — Directly Observed Therapy; Bipolar Disorder | interventions — Emotion-Focused Therapy; Psychotherapy

STUDY DESIGN:
Intervention Model Description: The research was designed as a single-blind randomized controlled trial (pre-test-post-test, control group, follow-up measurement) in an experimental setting.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group, where no intervention will be made and only research questionnaires will be applied (Placebo Comparator): The determined scale forms will be applied to the people in the control group who will be included in the study as a pre-test at the beginning of the study, as a post-test 10 days after the pre-test, and finally as a follow-up test one month after the pre-test.
  Interventions: Other: scale form
- intervention group to which emotion-focused therapy will be applied (Experimental): Participants in the intervention group will first be given face-to-face individual interviews to establish the therapeutic environment and relationship (Individual interviews are designed as orientation, diagnosis and planning stages, 30-minute interviews). Then, three intervention stages (40-minute, group therapy) will be applied and the last session will be both intervention (post-test application) and termination stage (completion of emotion-focused therapy application). After the individual interviews, individuals will be included in 3 intervention sessions as group training. It is planned that each group will have at least 4 and at most 6 people. If the specified number cannot be reached, the study will continue until the specified number is reached.
  Interventions: Other: Emotion Focused Therapy application; Other: scale form

INTERVENTIONS:
Other: Emotion Focused Therapy application — Participants in the intervention group will first be given face-to-face individual interviews to establish the therapeutic environment and relationship (Individual interviews are designed as orientation, diagnosis and planning stages, 30-minute interviews). Then, three intervention stages (40-minute, group therapy) will be applied and the last session will be both intervention (post-test application) and termination stage (completion of emotion-focused therapy application). After the individual interviews, individuals will be included in 3 intervention sessions as group training. It is planned that each group will have at least 4 and at most 6 people. If the specified number cannot be reached, the study will continue until the specified number is reached.
  Other Names: Emotion Focused Therapy; psychoeducation; psychotherapy
  Arms: intervention group to which emotion-focused therapy will be applied
Other: scale form — Emotion-focused therapy contributes to the treatment compliance and functionality of psychiatric patients.

SUMMARY:
4.503 / 5.000 Bipolar disorder is a serious mood disorder that requires lifelong treatment and is characterized by recurring periods of depression, mania, hypomania or mixed episodes without a specific order, completely normal between episodes or thought to be with minimal symptom levels, has a high mortality and morbidity rate, causes serious deterioration in the quality of life in terms of occupational, interpersonal, social, familial and economic aspects. It causes serious deterioration in the lives of patients due to suicide attempts, substance abuse, poor functionality, low academic success, deterioration in interpersonal communication and repeated hospitalizations. One of the conditions that most affects the course of the disease in bipolar disorder and causes recurrences is treatment compliance. Treatment compliance includes individuals accepting and applying the treatments recommended for their illness, going to check-ups, controlling their emotions, continuing treatment programs, using medications as often and at the dose prescribed, continuing other treatment methods and healthy behavioral changes (individual coping strategies, skills training, emotion management training, awareness training, etc.). In bipolar patients, where mood swings are frequent, emotional reactivity is one of the important factors affecting the treatment compliance process. The concept of emotional reactivity can be defined as the emotional sensitivity experienced by the individual in response to many stimuli and stimuli, the emotional intensity experienced strongly, and the emotional resistance shown during the period until reaching the basic emotion. The emotions that usually create emotional reactions are emotions such as anger, anxiety, stress, and hurt. Even individuals without a psychiatric diagnosis can sometimes have difficulty controlling such emotions when they encounter them. Therefore, it is very important for these bipolar individuals to have mood awareness so that they can recognize these emotions and exhibit appropriate behaviors towards emotions. Since individuals who are aware of their emotions will increase their emotional attention and emotional clarity, it becomes easier for them to recognize their emotions. Patients' compliance with treatment positively affects the course of the disease and supports the increase in functionality with regular treatment. Psychosocial interventions for patients with bipolar disorder contribute to a decrease in patients' symptoms, increased compliance with medical treatment, and a decrease in the need for rehospitalization, as well as increased social and occupational functioning. This study was planned to examine the effects of emotion-focused therapy applied to patients with bipolar disorder on the patients' mood awareness and emotional reactivity. The application of the study will be carried out with patients diagnosed with bipolar disorder in remission at the Psychiatry Clinic of Muğla Sıtkı Koçman University Faculty of Medicine Hospital after obtaining permissions. In determining the hospital where the study will be conducted, the current number of patients, accessibility, cooperation of the team, and the absence of structured group emotion-focused therapy studies in the institution were taken into consideration. The content of the emotion-focused therapy program planned to be used in the study was prepared by obtaining the opinions of expert faculty members working in different universities. The study was planned with bipolar disorder patients who were hospitalized in a psychiatric clinic and started the treatment process, and in an experimental setting (pre-test-post-test control group, follow-up measurement), 6 sessions were planned for the intervention group during their hospitalization, 2 days a week, the first 3 sessions were 30 minutes and the other 3 sessions were 40 minutes. Before starting the emotion-focused therapy, the purpose of the study was explained to the intervention group, the data collection tools were introduced, and their verbal and written permissions were obtained, and the pre-test was applied face to face. Face-to-face interviews and 6 sessions of emotion-focused therapy application will be held in the psychiatric clinic interview room. As the final test application, the scales will be applied face to face by the clinic nurse immediately after the last session of emotion-focused therapy. A follow-up test will be performed on the patients one month later. The patient will be met with a total of 7 times. It is assumed that the emotion-focused therapy application will increase the patient's ability to recognize individual emotions, manage emotions, medication compliance and functionality level after discharge.

DETAILED DESCRIPTION:
Bipolar disorder is defined as a mental disorder characterized by depression, hypomania, and manic episodes, regardless of order, with periods of remission between these episodes or where the symptoms are thought to be felt at very mild levels, requiring regular follow-up and treatment, and causing serious impairments in family, interpersonal, and occupational functioning (Yeloğlu & Hocaoğlu, 2017; Jung et al, 2020). The World Health Organization (WHO) has reported bipolar disorder as one of the top 10 diseases that cause disability among all diseases. Treatment compliance rates in bipolar disorder vary between 20% and 60%. The average prevalence rate of non-adherence to treatment is 41% (Zhang, 2020). The exact cause of this disease, which is known to cause high mortality and morbidity, has been associated with biological and psychosocial factors (Öztürk, 2020). This disorder is classified as subtypes under the title of "Bipolar Disorder and Related Disorders" in the "Diagnostic and Statistical Manual of Mental Disorders/DSM-5". These classifications are as follows; bipolar disorder I, bipolar disorder II, cyclothymia disorder, substance/medication-induced bipolar and related disorder, other specified and not otherwise specified bipolar and related disorder (Atagün & Oral, 2021). When all bipolar disorders are taken into account, it has been reported that the lifetime prevalence is approximately 7.8%. In order to prevent the recurrence of bipolar disorder, providing patients with functionality, improving their compliance with treatment and quality of life, and providing them with stress coping skills are among the most important goals of treatment (Özdel et al., 2021). Patients may experience serious disruptions in their lives due to suicide attempts, substance abuse, poor functionality, decreased academic success, poor interpersonal communication, and repeated hospitalizations. One of the conditions that most affects the course of the disease in bipolar disorder and causes relapses is treatment compliance. Treatment compliance includes individuals accepting and implementing the recommended treatments for their illness, going to check-ups, controlling their emotions, continuing treatment programs, using medications as often and at the dose they are prescribed, participating in psychosocial support treatment methods applied in addition to pharmacotherapy and making healthy behavioral changes (individual coping strategies, skills training, emotional management training, awareness training, etc.) (Moreira et al., 2017).

Emotional reactivity is one of the important factors affecting the treatment compliance process in bipolar patients, where mood swings are frequent (Miller & Black, 2020). The concept of emotional reactivity can be defined as the emotional sensitivity experienced by the individual in response to many stimuli and stimuli, the emotional intensity experienced strongly, and the emotional endurance shown until reaching the basic emotion (Seçer et al., 2013). Emotions that usually create emotional reactions are emotions such as anger, anxiety, stress, and hurt (Du et al., 2018). Even individuals without a psychiatric diagnosis can sometimes have difficulty controlling such emotions when they encounter them (Demissie et al., 2018). Therefore, it is very important for these bipolar individuals to have mood awareness so that they can recognize these emotions and exhibit appropriate behaviors towards emotions. Individuals who are aware of their emotions can have an easier time recognizing their emotions, as their emotional attention and emotional clarity will increase (Gökdağ & Yüvrük, 2022). Patients' compliance with treatment positively affects the course of the disease and supports increased functionality with regular treatment. Psychosocial interventions for patients with bipolar disorder contribute to a decrease in patients' symptoms, increased compliance with medical treatment, and a decrease in the need for rehospitalization, as well as increased social and occupational functionality (Subic-Wrana et al., 2014; Miziou et al., 2015). Studies have also shown that providing patients with psychosocial interventions aimed at understanding their emotions is important for increasing the effectiveness of bipolar disorder treatment and for the disease process to progress positively (Watson & Dodd, 2017). Emotion-focused therapy, which is among the interventions that can be applied, is an intervention strategy based on patients' recognition of emotions, development of emotional awareness and understanding, early detection of warning signs and mood changes, increasing compliance with treatment, and providing information about the disease (Demissie et al., 2018). Emotion-focused therapy (EFT) is a psychotherapy method based on the emotion-centered humanistic approach theory, which processes the awareness of emotions, acceptance, expression, regulation and transformation of emotions in the therapeutic process (Morriss et al., 2016). Thanks to the given emotion-focused therapy, individuals can gain awareness about their emotions and increase their functionality by developing individual skills in directing their reactions (Çam, & Çuhadar, 2013). Another therapy that is at the forefront of the theories that constitute the theoretical framework of DOT is the person-centered theory. According to this theory, the cause of psychological problems arises from the inconsistency between the individual's "self-concept" and "experience". When the inconsistency between the self-concept (I am strong) and experience (feeling weak) prevents awareness, the person reacts to this by worrying. Again, according to this theory, when the individual is guided by "self-actualization", which is the most basic tendency of human life, the person becomes reliable, believable and constructive. DOT argues that emotional change should be placed at the center of therapy in order to achieve permanent change and therefore adopts the modern emotion theory (Uslu & Gizir 2019). DOT suggests that emotions have an adaptive potential on their own if activated, and adopts the view that emotions help clients reorganize their negative self-experiences and change problematic emotional states and interactions. The main purpose of DOT is to strengthen the self, regulate affect, and create new meanings (Greenberg, 2016). Since there is no standardized emotion-focused therapy application that can be applied to patients with bipolar disorder in psychiatric clinics, it is thought that a well-designed therapy application can increase compliance with treatment and increase the level of functionality, thus maintaining the well-being of patients and reducing health care costs. This study was planned to examine the effect of emotion-focused therapy applied to patients with bipolar diagnosis on the patients' mood awareness and emotional reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria are being between the ages of 18-65,
2. Being diagnosed with Bipolar Disorder (I, II) and receiving maintenance treatment and being in remission,
3. Receiving standard drug treatment (mood stabilizer, antipsychotic or antidepressant) and standard clinical follow-up for bipolar disorder,
4. Not having hearing, comprehension and vision problems,
5. Being able to read and write,
6. Being patients who agree to participate in the study.

Exclusion Criteria:

1. Having another psychotic disorder in addition to the diagnosis of bipolar disorder,
2. Being newly diagnosed with bipolar disorder and being in the acute phase,
3. Wanting to leave the study,
4. Not agreeing to participate in the study,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
EFFECTS OF EMOTION-FOCUSED THERAPY APPLIED TO PATIENTS WITH BIPOLAR DIAGNOSIS ON THEIR MOOD AWARENESS AND EMOTIONAL REACTIVITY | 6 month
  By creating randomized controlled groups, emotion-focused therapy will be applied between the control and intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Eğitim Ve Araştırma Hastanesi, Multiple Locations, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shahar B. New Developments in Emotion-Focused Therapy for Social Anxiety Disorder. J Clin Med. 2020 Sep 10;9(9):2918. doi: 10.3390/jcm9092918. PMID 32927706
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32927706/